CLINICAL TRIAL: NCT06284317
Title: An International, Multicentre, Open-label Randomised Phase III Trial to Evaluate the Benefit of Adding Adjuvant Durvalumab After Neoadjuvant Chemotherapy Plus Durvalumab in Patients With Stage IIB-IIIB (N2) Resectable NSCLC
Brief Title: A Study to Evaluate the Benefit of Adding Durvalumab After Chemotherapy, Durvalumab and Surgery in Patients With Early-stage, Operable, Non-small Cell Lung Cancer.
Acronym: ADOPT-lung
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 25-23
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: IIB-IIIB (N2) resectable NSCLC; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): Protocol treatment in the adjuvant phase consists of adjuvant durvalumab
  Interventions: Drug: Adjuvant durvalumab
- Observation (No Intervention): Observation only

INTERVENTIONS:
Drug: Adjuvant durvalumab — Durvalumab is given at a fixed dose of 1500 mg i.v. every 4 weeks (±1 week) until relapse or unacceptable toxicity, for a maximum of 12 cycles after surgery.
  Arms: Durvalumab

SUMMARY:
ADOPT-lung is an international, multicentre, open-label randomised phase III trial. Protocol treatment consists of 3-4 cycles of neoadjuvant durvalumab in combination with platinum-based doublet chemotherapy, followed by surgery. Patients with R0 and R1 only resection will be randomised to receive either adjuvant durvalumab for 12 cycles (experimental arm) or observation (control arm). The primary objective of the study is to determine whether additional adjuvant immunotherapy with durvalumab after neoadjuvant chemo-immunotherapy has an effect on disease-free survival (DFS) in patients who do not achieve complete pathological response (pCR) as per local assessment according to the IASLC recommendations.

ELIGIBILITY:
Inclusion Criteria for enrolment:

* Histologically confirmed NSCLC.
* Stage IIB-IIIB (T1-4 N0-2) according to 8th edition of the TNM staging system of lung cancer.

Stage III assessment should include samples of lymph nodes at levels 4, bilaterally, and level 7 to rule out stage IIIB N3 disease.

T4 tumours will only be eligible if they are defined as T4 based only on their size (>7cm); any other reason will be considered ineligible.

* Known PD-L1 status, as tested locally using a validated assay. To ensure comparability of results, it is strongly encouraged that PD-L1 testing is done with the Ventana PD-L1 (SP263) assay.
* Absence of EGFR mutation or ALK translocation, as tested locally.
* Primary tumour resectable and functionally operable as assessed per local multidisciplinary tumour board (cardiac evaluation, pulmonary function and diffusion capacity, comorbidity).
* Adequate haematological function:

Haemoglobin ≥90 g/L, Absolute neutrophil count (ANC) ≥1.0× 109/L, Platelet count ≥75× 109/L.

- Adequate renal function: Measured creatinine clearance (CL) >40 mL/min or calculated CL >40 mL/min calculated by the Cockcroft-Gault.

- Adequate liver function: ALT and AST ≤2.5× institutional ULN, Total serum bilirubin ≤1.5× institutional ULN (patients with Gilbert's syndrome may be allowed to be enrolled after consultation with the Medical Affairs Team at the ETOP IBCSG Partners Foundation.

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Age ≥18 at the time of enrolment.
* Body weight >30 kg.
* Life expectancy of at least 12 weeks.
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test at screening before enrolment. Pregnancy test must be repeated within 3 days before the first dose of protocol treatment.
* Written IC for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention.

Eligibility Criteria for randomisation:

* Surgical resection must have been completed. Note: Participants who have had only had segmentectomy or wedge resections are not eligible for randomisation.
* Patients must have complete resection: R0 or R1 resection.
* Patients must be fit to receive adjuvant treatment with durvalumab.
* Patients must have no evidence of metastatic disease as assessed by CT scan.
* Documentation of pathological response as per local review must be available.

Exclusion Criteria for enrolment:

* T4 with invasion of heart, great vessels, carina, trachea, oesophagus, or spine.
* Any previous or concurrent treatments for NSCLC.
* Any previous immunotherapy.
* Major surgical procedure (as per investigators assessment) within 28 days before enrolment.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune disease or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

Patients with vitiligo or alopecia. Patients with type I diabetes. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.

Any chronic skin condition that does not require systemic therapy. Patients without active disease in the last 5 years may be included but only after consultation with the Medical Affairs Team at the ETOP IBCSG Partners Foundation.

Patients with celiac disease controlled by diet alone.

* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease (ILD), or serious chronic gastrointestinal conditions associated with diarrhoea.
* Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of another primary malignancy except for:

Malignancy treated with curative-intent and with no known active disease 5 years before the first dose of durvalumab and of low potential risk for recurrence.

Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.

Adequately treated carcinoma in situ without evidence of disease.

* History of leptomeningeal carcinomatosis.
* History of active primary immunodeficiency.
* Active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HbsAg) or HBV core antibody (anti-HBc).

Participants with a past or resolved HBV infection (defined as the presence of anti-HBc and absence of HbsAg) are eligible.

Participants positive for HCV antibody are only eligible if polymerase chain reaction is negative for HCV RNA.

* Known HIV infection that is not well-controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load for 3 months, CD4+ count of 500 cell per mm3, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 3 months on the same anti-HIV medication.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).

Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or its equivalent.

Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).

- Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab.

Note: Patients in the ADOPT-lung trial, should not receive live vaccine whilst receiving durvalumab and for up to 30 days after the last dose.

Concurrent enrolment in another interventional clinical trial.

* Known allergy or suspected hypersensitivity to durvalumab or its excipients.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Female patients who are pregnant or in the period of lactation.
* Female patients of childbearing potential and sexually active men who are not willing to use a highly effective contraceptive method during the trial until at least 90 days after the last dose of protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase.
  DFS is defined as the time from the date of randomisation until disease recurrence (including loco-regional recurrence, a distant (metastatic) recurrence or a second primary) or death from any cause. Censoring (for patients without recurrence/death) will occur at the date of last tumour assessment. Patients without a post-randomisation tumour assessment will be censored at the date of randomisation (plus 1 day). DFS will be assessed in patients without pCR (primary endpoint), as well as in patients with pCR (secondary endpoint) and in patients with/without ctDNA clearance (secondary endpoints).

SECONDARY OUTCOMES:
DFS in patients with pCR | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase (after randomisation).
  DFS is defined as the time from the date of randomisation until disease recurrence (including loco-regional recurrence, a distant (metastatic) recurrence or a second primary) or death from any cause. Censoring (for patients without recurrence/death) will occur at the date of last tumour assessment. Patients without a post-randomisation tumour assessment will be censored at the date of randomisation (plus 1 day). DFS will be assessed in patients without pCR (primary endpoint), as well as in patients with pCR (secondary endpoint) and in patients with/without ctDNA clearance (secondary endpoints).
Overall survival (OS) in patients with/without pCR | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase (after randomisation).
  OS is defined as the time from the date of randomisation until death from any cause. Censoring (for patients who are not reported as having died) will occur at the date when they were last known to be alive. Patients without post-randomisation information will be censored at the date of randomisation (plus 1 day). OS will be assessed in patients with/without pCR.
DFS in patients with/without ctDNA clearance | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase (after randomisation).
Time to recurrence (TTR) in patients with/without pCR | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase (after randomisation).
  TTR is defined as the time from the date of randomisation until disease recurrence. Censoring (for patients without recurrence) will occur at the date of the last tumour assessment. Patients without a post-randomisation tumour assessment will be censored at the date of randomisation (plus 1 day). TTR will be assessed in patients with/without pCR.
Time to treatment discontinuation (TTD) in patients with/without pCR | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase (after randomisation).
Toxicity according to CTCAE v5.0 | From the date of randomisation until last patient last visit (approximately 60 months after randomisation of the first patient)
  Assessed in the adjuvant treatment phase (after randomisation).
  All safety parameters will be summarised in tables to evaluate the toxicity/safety profile of the protocol treatment based on:
  * Adverse events according to CTCAE v5.0 (any-cause as well as treatment-related) including adverse events leading to dose interruptions, withdrawal of protocol treatment, and death.
  * Severe, serious, and selected adverse events.
  * Deaths.
  * Laboratory parameters and abnormalities, and vital signs.

OTHER OUTCOMES:
Correlation between ctDNA clearance and DFS | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  Exploratory endpoint
Correlation between ctDNA clearance and OS | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  Exploratory endpoint
Correlation between ctDNA clearance and initial PD-L1 assessment | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  Exploratory endpoint
Outcome (event-free survival) | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  Outcome (EFS) in patients with patients with either
  * ctDNA clearance after neoadjuvant treatment but not achieving pCR
  * no ctDNA clearance after neoadjuvant treatment but achieving pCR
Correlation of Outcome Disease-free survival (DFS) | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  Correlation of Outcome (DFS) in patients with longitudinal ctDNA assessment
Correlation of Outcome Overall survival (OS) | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  Correlation of Outcome (OS) in patients with longitudinal ctDNA assessment
pCRDescription of patients entering each phase (e.g., % surgery, % randomised) | From the date of screening until last patient last visit (approximately 60 months after randomisation of the first patient)
  pCRDescription of patients entering each phase (e.g., % surgery, % randomised)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD-PhD, Study Chair — Centre Hospitalier Universitaire Vaudois, 1011 Lausanne, Switzerland; Sabine Schmid, MD, Study Chair — Inselspital, Universitätsspital Bern, 3010 Bern, Switzerland; Paul Van Schil, MD-PhD, Study Chair — Antwerp University Hospital, Antwerp, Belgium,; Stephen Finn, MD-PhD, Study Chair — St. James's Hospital, Dublin 8, Ireland
Locations (42):
- Australia (10):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Eastern Health, Box Hill, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Wien AKH, Vienna, Austria
- Belgium (2):
  - Institut Jules Bordet - HUB, Anderlecht
  - Antwerp University Hospital, Antwerp
- North Estonia Medical Centre Foundation, Talinn, Estonia
- France (4):
  - CHU Angers, Angers
  - Institut Bergonié, Bordeaux
  - Le Mans - CHG, Le Mans
  - Lyon - Centre Léon Bérard, Lyon
- Ireland (2):
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
- Italy (6):
  - SS Antonio e Biagio e Cesare Arrigo Hospital, Alessandria
  - Istituto Oncologico Veneto, Padua
  - Perugia Hospital, Perugia
  - Istituto Nazionale Tumori "Regina Elena", Rome
  - AOUS Policlinico Le Scotte, Siena
  - Universita di Verona - Department of Medicine, Verona
- Netherlands (2):
  - NKI, Amsterdam
  - UMCU, Utrecht
- Switzerland (9):
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Eoc - Iosi, Bellinzona
  - Inselspital Bern, Bern
  - HFR Hôpital Fribourgeois, Fribourg
  - CHUV, Lausanne
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - University Hospital Zurich, Zurich
- United Kingdom (5):
  - Barts Health NHS Trust, London
  - Royal Marsden Hospital (Chelsea), London
  - Royal Marsden Hospital (Sutton), London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester